CLINICAL TRIAL: NCT07173842
Title: Establishment of the NeuroPsyBiT-BD Omics Program: Development of a Turkish Bipolar Disorder Biobank Integrating Genomic and Epigenomic Profiling With Structured Clinical Phenotyping and Secure Data Infrastructure
Brief Title: NeuroPsyBiT-BD Omics: Genomic & Epigenomic Biobank of Bipolar Disorder
Acronym: NeuroPsyBiT-BD
Status: Not yet recruiting | Type: Observational
Sponsor: Selçuk State Hospital (Other)
Collaborators: Research and Treatment Society of Genetic Disorders (Other)
Responsible Party: Principal Investigator, Rukiye Tekdemir, Associate Professor Dr., Selçuk State Hospital
Other Study IDs: NEUROPSYBIT-BD-001; TÜBİTAK 1505 (Other: TÜBİTAK 1505 University-Industry Collaboration Application); RTSGD-BD-BIOBANK-2025 (Other: RTSGD Internal Project Code); to be updated after approval (Other: Selçuk University Medical Faculty Ethics Committee Reference Number)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Mood Disorders; Psychiatric Genetics; Epigenomics; GWAS; EWAS; Biobank; Phenotyping
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected in EDTA tubes from individuals diagnosed with bipolar disorder. DNA will be extracted from these samples for use in genomic and epigenomic analyses, including genome-wide association studies (GWAS) and epigenome-wide association studies (EWAS). Plasma and buffy coat fractions may also be stored for future biomarker studies. All biospecimens will be processed and stored under ISO-compliant biobanking standards with barcode tracking to ensure quality, traceability, and secure long-term retention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bipolar Disorder Patients: Participants clinically diagnosed with bipolar disorder, recruited under ethics committee-approved protocols. Detailed phenotypic, clinical, and psychosocial parameters will be collected using the NeuroCybe Data Collector system. Biospecimens (e.g., EDTA blood samples) will be stored in the RTSGD-NeuroPsyBiT Biobank under ISO-compliant standards.
  Interventions: Other: Biobanking and Phenotypic Data Collection
- Control Group: Healthy volunteers without a history of psychiatric disorders, matched for key demographic variables (age, sex). Biospecimens and phenotypic data will be collected following the same standardized procedures as the patient cohort. Controls provide baseline references for genomic, epigenomic, and phenotypic comparisons.
  Interventions: Other: Biobanking and Phenotypic Data Collection

INTERVENTIONS:
Other: Biobanking and Phenotypic Data Collection — This intervention involves the systematic collection of blood samples (EDTA tubes for DNA extraction) and detailed phenotypic/clinical data using the NeuroCybe Data Collector software. All biospecimens are processed and stored at the RTSGD-NeuroPsyBiT Biobank under ISO-compliant procedures. Data are entered into a secure on-premises server infrastructure (GDPR/KVKK compliant) for long-term use in genomic and epigenomic studies. No therapeutic intervention is applied; all activities are non-invasive and focused on sample and data acquisition.

SUMMARY:
Brief Summary The goal of this observational study is to establish a comprehensive biobank and phenotypic data repository for patients diagnosed with bipolar disorder in Türkiye. The study will prospectively collect standardized clinical, demographic, lifestyle, and biological data to create a secure genomic and epigenomic research resource.

The main questions it aims to answer are:

Can large-scale, standardized phenotypic and biological data collection improve the understanding of bipolar disorder subtypes and disease course?

Can integration of biobank samples with genomic and epigenomic analyses identify biomarkers that inform future diagnosis, prognosis, and treatment strategies?

Participants will:

Provide consent and demographic/clinical information using the NeuroPsyBiT Data Collector software.

Contribute blood samples (e.g., EDTA tubes) for DNA extraction, genotyping, and future epigenomic studies.

Allow secure storage of their data and biospecimens in the RTSGD biobank for use in ethically approved research projects.

All data and samples will be collected and stored under strict ethical oversight and in compliance with national (KVKK) and international (GDPR) data protection regulations. Personally identifiable information will not be shared, and access to the biobank and dataset will only be granted after approval by institutional review boards and ethics committees.

This registry will create the foundation for future genome-wide association studies (GWAS) and epigenome-wide association studies (EWAS), supporting the long-term goal of developing precision psychiatry tools for bipolar disorder.

DETAILED DESCRIPTION:
This project, NeuroPsyBiT-BD-001: Genomic & Epigenomic Biobank of Bipolar Disorder, is an observational patient registry designed to establish a large-scale biobank and standardized phenotypic data platform for individuals with bipolar disorder in Türkiye.

Objectives and Rationale:

Bipolar disorder (BD) is a chronic and heterogeneous psychiatric condition with high morbidity, relapse rates, and unmet clinical needs. Genetic and epigenetic factors are believed to play a central role in its pathogenesis, yet reliable biomarkers remain scarce. By combining deeply phenotyped clinical data with biological samples, this registry seeks to create a robust foundation for genome-wide association studies (GWAS) and epigenome-wide association studies (EWAS). This approach will enable future biomarker discovery, stratification of subtypes, and exploration of treatment response predictors.

Study Design:

Population: Patients diagnosed with bipolar disorder according to DSM-5 criteria will be recruited through the NeuroPsyBiT consortium, a partnership between the Research and Treatment Society of Genetic Disorders (RTSGD) and the Department of Psychiatry at Selçuk University Medical Faculty.

Sample Size: The initial target is 500 patients in the first phase, with an expansion goal of ≥1,000 patients within one year.

Data Collection: Phenotypic and clinical data (>250 variables) will be systematically recorded using the NeuroCybe Data Collector, a proprietary software platform developed for standardized psychiatric data capture. Domains include demographics, medical/psychiatric history, clinical course, comorbidities, lifestyle/exposome, treatments, and psychometric assessments.

Biospecimen Collection: Blood samples (EDTA tubes) will be collected for DNA extraction, genotyping, and future methylation profiling. Samples will be processed and stored under ISO-compliant biobanking standards, ensuring traceability and long-term integrity.

Infrastructure and Data Security:

Biobank Management: RTSGD laboratories will serve as the central biobank facility, operating under internationally recognized quality standards for sample processing and storage.

Data Governance: All phenotypic and genotypic data will be securely stored on RTSGD on-premise servers with no cloud storage permitted.

Ethics & Privacy: Data handling will strictly comply with national (KVKK) and international (GDPR) regulations. Personally identifiable information will be de-identified. Data access will only be granted following approval by both institutional ethics committees and the Turkish Ministry of Health.

Future Access: De-identified datasets and biospecimens will be made available for national and international collaboration upon direct application to the consortium, subject to ethical approvals.

Scientific Impact:

This registry represents the first large-scale, ISO-standardized biobank for bipolar disorder in Türkiye. By unifying deep phenotyping with genomic and epigenomic resources, it will:

Enable high-resolution GWAS and EWAS in BD.

Provide a resource for cross-cohort meta-analysis and replication studies.

Facilitate translational research toward precision psychiatry approaches (diagnostic tools, risk stratification, and individualized treatment).

Create a sustainable national and international platform for collaboration in psychiatric genetics and epigenetics.

Long-term Vision:

The NeuroPsyBiT-BD registry is designed as a scalable infrastructure. In its initial phases, it will serve national research priorities; over time, it will expand to international collaborations, training opportunities, and joint projects. By combining phenotypic richness with state-of-the-art genomic technologies, the registry will contribute significantly to global efforts aimed at unraveling the biological basis of bipolar disorder.

ELIGIBILITY:
Inclusion Criteria (Bipolar Disorder Cohort):

* Age 18-65 years.
* DSM-5 diagnosis of Bipolar I, II and NOS confirmed by SCID-5.
* Able to provide written informed consent.
* Willing to complete standardized phenotyping (e.g., YMRS, HDRS-17, FAST/WHODAS) and to provide biospecimens (minimum: whole blood in EDTA; optional: serum, plasma, PAXgene-RNA, cfDNA tubes).
* Stable psychotropic regimen for ≥14 days prior to sampling or drug-free for ≥14 days.

Inclusion Criteria (Control Cohort):

* Age 18-65 years.
* No lifetime DSM-5 psychiatric disorder (including bipolar and schizophrenia spectrum and others) by SCID-5.
* No first-degree family history of major psychiatric disorder (including bipolar and schizophrenia spectrum).
* Able to provide informed consent and blood samples for biobanking.
* No current psychotropic medication.

Exclusion Criteria (applies to both cohorts):

* Presence of neurological disorders (e.g., epilepsy, multiple sclerosis, Parkinson's disease).
* Severe, uncontrolled medical illness that could affect participation or biological measures (e.g., decompensated cardiac, renal, hepatic, or endocrine disease).
* Active infection or fever within 14 days; systemic corticosteroids or immunomodulators within 30 days; vaccination within 14 days.
* Blood transfusion within 3 months or blood donation within 2 weeks prior to sampling.
* Current substance use disorder.
* Pregnancy or breastfeeding at enrollment.
* Inability to comply with procedures or lack of capacity to consent (e.g., significant cognitive impairment, severe language barrier), or acute mania/psychosis requiring immediate hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited through the Department of Psychiatry at Selçuk University Medical Faculty in Konya, Türkiye, in collaboration with the Research and Treatment Society of Genetic Disorders (RTSGD) and the NeuroPsyBiT Consortium. The population includes adults aged 18-65 diagnosed with bipolar disorder who receive outpatient or inpatient psychiatric care at Selçuk University clinical facilities, as well as healthy control volunteers recruited from the local community and hospital staff. Both patient and control groups will contribute to the establishment of a national biobank and phenotypic data registry designed to support future genomic and epigenomic studies
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Successfully Collected and Biobanked DNA Samples | From enrollment to 24 months
  Count of bipolar disorder participants whose blood samples (EDTA tubes) are successfully collected, processed, quality-checked (DNA yield/purity), and stored in the RTSGD-NeuroPsyBiT Biobank under ISO standards

SECONDARY OUTCOMES:
Completeness of Phenotypic Dataset per Participant | 24 months
  Proportion of participants with ≥95% of required variables (demographics, psychiatric history, medication, psychometric scales, metabolic markers, family history) successfully collected via the NeuroCybe Data Collector system.
Proportion of Biobanked Samples Ready for Genomic/Epigenomic Analysis | 24 months
  Proportion of stored samples that meet Illumina Infinium platform quality thresholds (DNA concentration, integrity, and QC metrics) for downstream GWAS/EWAS.
Rate of Successful Data-Sample Linkage | 24 months
  Percentage of participants whose biospecimens are securely linked to their clinical and phenotypic data in the RTSGD on-premises server system, validated by barcoding and audit trail.

CONTACTS AND LOCATIONS:
Locations (1):
- Selçuk University Faculty of Medicine, Department of Psychiatry / NeuroPsyBiT-RTSGD Consortium, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified (pseudonymised) IPD will be shared for verification/secondary/meta-research under controlled access, per FAIR+GDPR; minimal. Sociodemographics: age (bands), sex/gender, marital, education, SES/employment, region; gravidity/miscarriages; ethnicity where permitted. Clinical: onset age; prior psychiatric history; episode #/polarity; mixed/rapid-cycling/psychosis; hospitalisations; treatment history (dose/duration/levels); family history; suicidality; comorbidities; concomitant meds. Scales: HDRS/HAM-D, YMRS, ALDA, CGI, UKU, FAST, WHOQOL-BREF-TR, PSQI, MEQ-SF, MCTQ, CTQ-53, ASRS, SPS. Lifestyle: tobacco, alcohol, illicit, caffeine; sleep-wake regularity. Labs/biometrics: metabolic-syndrome, BMI, renal/liver, electrolytes, ESR/routine, HR, ECG; QRISK3 (derived score+timepoint only). Biospecimen metadata: type, timepoint, processing, storage, QC; no primary specimens or genomic raw data without approval. Docs: data dictionary/codebook, CRFs, scoring refs, derivation readme.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Individual Participant Data (IPD) and supporting documentation (Study Protocol, SAP, ICF, Analytic Code) will become available 12 months after study completion and will remain accessible for 5 years under controlled access agreements. After this period, renewal of access may be possible upon approval by the sponsor and the Turkish Health Ministry.
Access Criteria: Only qualified researchers affiliated with recognized academic or clinical institutions may apply.
  Requests must be accompanied by a formal research proposal, including clear objectives, methodology, and justification for data use.
  All requests require Ethics Committee approval and explicit authorization from the Turkish Ministry of Health.
  Data will be shared only in a de-identified, encrypted format via a secure on-premises or ministry-approved platform. No direct downloads or cloud transfer will be allowed.
  Applicants must sign a Data Use Agreement (DUA), prohibiting re-identification attempts, redistribution, or secondary use beyond the approved proposal.
  Publication of analyses derived from the IPD will require pre-review by the sponsor consortium (RTSGD/NeuroPsyBiT) to ensure compliance with ethical, legal, and scientific standards.
  Violations of these criteria will result in immediate termination of access and legal consequences under Turkish data protection laws (KVKK) an
URL: https://www.neuropsybit.org/data-governance

REFERENCES:
- [Background] Marovic B, Curcin V. Impact of the European General Data Protection Regulation (GDPR) on Health Data Management in a European Union Candidate Country: A Case Study of Serbia. JMIR Med Inform. 2020 Apr 17;8(4):e14604. doi: 10.2196/14604. PMID 32301736
- [Background] Molnar-Gabor F, Beauvais MJS, Bernier A, Jimenez MPN, Recuero M, Knoppers BM. Bridging the European Data Sharing Divide in Genomic Science. J Med Internet Res. 2022 Oct 19;24(10):e37236. doi: 10.2196/37236. PMID 36260387
- [Background] Talu CK, Toper MH, Sahin Y, Erdogdu IH. Pathology and Biobanking. Turk Patoloji Derg. 2020;36(2):93-108. doi: 10.5146/tjpath.2020.01482. PMID 32189322
- [Background] Bernier A, Molnar-Gabor F, Knoppers BM, Borry P, Cesar PMDG, Devriendt T, Goisauf M, Murtagh M, Jimenez PN, Recuero M, Rial-Sebbag E, Shabani M, Wilson RC, Zaccagnini D, Maxwell L. Reconciling the biomedical data commons and the GDPR: three lessons from the EUCAN ELSI collaboratory. Eur J Hum Genet. 2024 Jan;32(1):69-76. doi: 10.1038/s41431-023-01403-y. Epub 2023 Jun 15. PMID 37322132
- [Background] Owusu SA. Ethical implications of the widespread use of informal mHealth methods in Ghana. J Med Ethics. 2024 Jul 23;50(8):563-568. doi: 10.1136/medethics-2021-107920. PMID 35396337
- [Background] Yakubu A, Munung NS, De Vries J. How Should Biobanking Be Governed in Low-Resource Settings? AMA J Ethics. 2020 Feb 1;22(2):E156-163. doi: 10.1001/amajethics.2020.156. PMID 32048586
- [Background] Kilkku N, Halkoaho A. Informed consent, genomic research and mental health: A integrative review. Nurs Ethics. 2022 Jun;29(4):973-987. doi: 10.1177/09697330211066573. Epub 2022 Feb 4. PMID 35119339
- [Background] Campbell LD, Astrin JJ, DeSouza Y, Giri J, Patel AA, Rawley-Payne M, Rush A, Sieffert N. The 2018 Revision of the ISBER Best Practices: Summary of Changes and the Editorial Team's Development Process. Biopreserv Biobank. 2018 Feb;16(1):3-6. doi: 10.1089/bio.2018.0001. Epub 2018 Feb 2. PMID 29393664
- [Background] Akyuz K, Goisauf M, Martin GM, Mayrhofer MT, Antoniou S, Charalambidou G, Deltas C, Malatras A, Papagregoriou G, Stefanou C, Voutounou M. Risk mapping for better governance in biobanking: the case of biobank.cy. Front Genet. 2024 Jun 14;15:1397156. doi: 10.3389/fgene.2024.1397156. eCollection 2024. PMID 38948356
- [Background] Ochang P, Stahl BC, Eke D. The ethical and legal landscape of brain data governance. PLoS One. 2022 Dec 29;17(12):e0273473. doi: 10.1371/journal.pone.0273473. eCollection 2022. PMID 36580464
- [Background] Eke DO, Bernard A, Bjaalie JG, Chavarriaga R, Hanakawa T, Hannan AJ, Hill SL, Martone ME, McMahon A, Ruebel O, Crook S, Thiels E, Pestilli F. International data governance for neuroscience. Neuron. 2022 Feb 16;110(4):600-612. doi: 10.1016/j.neuron.2021.11.017. Epub 2021 Dec 15. PMID 34914921
- [Background] Pisanu C, Meloni A, Severino G, Squassina A. Genetic and Epigenetic Markers of Lithium Response. Int J Mol Sci. 2022 Jan 29;23(3):1555. doi: 10.3390/ijms23031555. PMID 35163479
- [Background] Muneer A. The Discovery of Clinically Applicable Biomarkers for Bipolar Disorder: A Review of Candidate and Proteomic Approaches. Chonnam Med J. 2020 Sep;56(3):166-179. doi: 10.4068/cmj.2020.56.3.166. Epub 2020 Sep 24. PMID 33014755
- [Background] Legrand A, Iftimovici A, Khayachi A, Chaumette B. Epigenetics in bipolar disorder: a critical review of the literature. Psychiatr Genet. 2021 Feb 1;31(1):1-12. doi: 10.1097/YPG.0000000000000267. PMID 33290382
- [Background] Mullins N, Forstner AJ, O'Connell KS, Coombes B, Coleman JRI, Qiao Z, Als TD, Bigdeli TB, Borte S, Bryois J, Charney AW, Drange OK, Gandal MJ, Hagenaars SP, Ikeda M, Kamitaki N, Kim M, Krebs K, Panagiotaropoulou G, Schilder BM, Sloofman LG, Steinberg S, Trubetskoy V, Winsvold BS, Won HH, Abramova L, Adorjan K, Agerbo E, Al Eissa M, Albani D, Alliey-Rodriguez N, Anjorin A, Antilla V, Antoniou A, Awasthi S, Baek JH, Baekvad-Hansen M, Bass N, Bauer M, Beins EC, Bergen SE, Birner A, Bocker Pedersen C, Boen E, Boks MP, Bosch R, Brum M, Brumpton BM, Brunkhorst-Kanaan N, Budde M, Bybjerg-Grauholm J, Byerley W, Cairns M, Casas M, Cervantes P, Clarke TK, Cruceanu C, Cuellar-Barboza A, Cunningham J, Curtis D, Czerski PM, Dale AM, Dalkner N, David FS, Degenhardt F, Djurovic S, Dobbyn AL, Douzenis A, Elvsashagen T, Escott-Price V, Ferrier IN, Fiorentino A, Foroud TM, Forty L, Frank J, Frei O, Freimer NB, Frisen L, Gade K, Garnham J, Gelernter J, Giortz Pedersen M, Gizer IR, Gordon SD, Gordon-Smith K, Greenwood TA, Grove J, Guzman-Parra J, Ha K, Haraldsson M, Hautzinger M, Heilbronner U, Hellgren D, Herms S, Hoffmann P, Holmans PA, Huckins L, Jamain S, Johnson JS, Kalman JL, Kamatani Y, Kennedy JL, Kittel-Schneider S, Knowles JA, Kogevinas M, Koromina M, Kranz TM, Kranzler HR, Kubo M, Kupka R, Kushner SA, Lavebratt C, Lawrence J, Leber M, Lee HJ, Lee PH, Levy SE, Lewis C, Liao C, Lucae S, Lundberg M, MacIntyre DJ, Magnusson SH, Maier W, Maihofer A, Malaspina D, Maratou E, Martinsson L, Mattheisen M, McCarroll SA, McGregor NW, McGuffin P, McKay JD, Medeiros H, Medland SE, Millischer V, Montgomery GW, Moran JL, Morris DW, Muhleisen TW, O'Brien N, O'Donovan C, Olde Loohuis LM, Oruc L, Papiol S, Pardinas AF, Perry A, Pfennig A, Porichi E, Potash JB, Quested D, Raj T, Rapaport MH, DePaulo JR, Regeer EJ, Rice JP, Rivas F, Rivera M, Roth J, Roussos P, Ruderfer DM, Sanchez-Mora C, Schulte EC, Senner F, Sharp S, Shilling PD, Sigurdsson E, Sirignano L, Slaney C, Smeland OB, Smith DJ, Sobell JL, Soholm Hansen C, Soler Artigas M, Spijker AT, Stein DJ, Strauss JS, Swiatkowska B, Terao C, Thorgeirsson TE, Toma C, Tooney P, Tsermpini EE, Vawter MP, Vedder H, Walters JTR, Witt SH, Xi S, Xu W, Yang JMK, Young AH, Young H, Zandi PP, Zhou H, Zillich L; HUNT All-In Psychiatry; Adolfsson R, Agartz I, Alda M, Alfredsson L, Babadjanova G, Backlund L, Baune BT, Bellivier F, Bengesser S, Berrettini WH, Blackwood DHR, Boehnke M, Borglum AD, Breen G, Carr VJ, Catts S, Corvin A, Craddock N, Dannlowski U, Dikeos D, Esko T, Etain B, Ferentinos P, Frye M, Fullerton JM, Gawlik M, Gershon ES, Goes FS, Green MJ, Grigoroiu-Serbanescu M, Hauser J, Henskens F, Hillert J, Hong KS, Hougaard DM, Hultman CM, Hveem K, Iwata N, Jablensky AV, Jones I, Jones LA, Kahn RS, Kelsoe JR, Kirov G, Landen M, Leboyer M, Lewis CM, Li QS, Lissowska J, Lochner C, Loughland C, Martin NG, Mathews CA, Mayoral F, McElroy SL, McIntosh AM, McMahon FJ, Melle I, Michie P, Milani L, Mitchell PB, Morken G, Mors O, Mortensen PB, Mowry B, Muller-Myhsok B, Myers RM, Neale BM, Nievergelt CM, Nordentoft M, Nothen MM, O'Donovan MC, Oedegaard KJ, Olsson T, Owen MJ, Paciga SA, Pantelis C, Pato C, Pato MT, Patrinos GP, Perlis RH, Posthuma D, Ramos-Quiroga JA, Reif A, Reininghaus EZ, Ribases M, Rietschel M, Ripke S, Rouleau GA, Saito T, Schall U, Schalling M, Schofield PR, Schulze TG, Scott LJ, Scott RJ, Serretti A, Shannon Weickert C, Smoller JW, Stefansson H, Stefansson K, Stordal E, Streit F, Sullivan PF, Turecki G, Vaaler AE, Vieta E, Vincent JB, Waldman ID, Weickert TW, Werge T, Wray NR, Zwart JA, Biernacka JM, Nurnberger JI, Cichon S, Edenberg HJ, Stahl EA, McQuillin A, Di Florio A, Ophoff RA, Andreassen OA. Genome-wide association study of more than 40,000 bipolar disorder cases provides new insights into the underlying biology. Nat Genet. 2021 Jun;53(6):817-829. doi: 10.1038/s41588-021-00857-4. Epub 2021 May 17. PMID 34002096
- [Background] Stahl EA, Breen G, Forstner AJ, McQuillin A, Ripke S, Trubetskoy V, Mattheisen M, Wang Y, Coleman JRI, Gaspar HA, de Leeuw CA, Steinberg S, Pavlides JMW, Trzaskowski M, Byrne EM, Pers TH, Holmans PA, Richards AL, Abbott L, Agerbo E, Akil H, Albani D, Alliey-Rodriguez N, Als TD, Anjorin A, Antilla V, Awasthi S, Badner JA, Baekvad-Hansen M, Barchas JD, Bass N, Bauer M, Belliveau R, Bergen SE, Pedersen CB, Boen E, Boks MP, Boocock J, Budde M, Bunney W, Burmeister M, Bybjerg-Grauholm J, Byerley W, Casas M, Cerrato F, Cervantes P, Chambert K, Charney AW, Chen D, Churchhouse C, Clarke TK, Coryell W, Craig DW, Cruceanu C, Curtis D, Czerski PM, Dale AM, de Jong S, Degenhardt F, Del-Favero J, DePaulo JR, Djurovic S, Dobbyn AL, Dumont A, Elvsashagen T, Escott-Price V, Fan CC, Fischer SB, Flickinger M, Foroud TM, Forty L, Frank J, Fraser C, Freimer NB, Frisen L, Gade K, Gage D, Garnham J, Giambartolomei C, Pedersen MG, Goldstein J, Gordon SD, Gordon-Smith K, Green EK, Green MJ, Greenwood TA, Grove J, Guan W, Guzman-Parra J, Hamshere ML, Hautzinger M, Heilbronner U, Herms S, Hipolito M, Hoffmann P, Holland D, Huckins L, Jamain S, Johnson JS, Jureus A, Kandaswamy R, Karlsson R, Kennedy JL, Kittel-Schneider S, Knowles JA, Kogevinas M, Koller AC, Kupka R, Lavebratt C, Lawrence J, Lawson WB, Leber M, Lee PH, Levy SE, Li JZ, Liu C, Lucae S, Maaser A, MacIntyre DJ, Mahon PB, Maier W, Martinsson L, McCarroll S, McGuffin P, McInnis MG, McKay JD, Medeiros H, Medland SE, Meng F, Milani L, Montgomery GW, Morris DW, Muhleisen TW, Mullins N, Nguyen H, Nievergelt CM, Adolfsson AN, Nwulia EA, O'Donovan C, Loohuis LMO, Ori APS, Oruc L, Osby U, Perlis RH, Perry A, Pfennig A, Potash JB, Purcell SM, Regeer EJ, Reif A, Reinbold CS, Rice JP, Rivas F, Rivera M, Roussos P, Ruderfer DM, Ryu E, Sanchez-Mora C, Schatzberg AF, Scheftner WA, Schork NJ, Shannon Weickert C, Shehktman T, Shilling PD, Sigurdsson E, Slaney C, Smeland OB, Sobell JL, Soholm Hansen C, Spijker AT, St Clair D, Steffens M, Strauss JS, Streit F, Strohmaier J, Szelinger S, Thompson RC, Thorgeirsson TE, Treutlein J, Vedder H, Wang W, Watson SJ, Weickert TW, Witt SH, Xi S, Xu W, Young AH, Zandi P, Zhang P, Zollner S; eQTLGen Consortium; BIOS Consortium; Adolfsson R, Agartz I, Alda M, Backlund L, Baune BT, Bellivier F, Berrettini WH, Biernacka JM, Blackwood DHR, Boehnke M, Borglum AD, Corvin A, Craddock N, Daly MJ, Dannlowski U, Esko T, Etain B, Frye M, Fullerton JM, Gershon ES, Gill M, Goes F, Grigoroiu-Serbanescu M, Hauser J, Hougaard DM, Hultman CM, Jones I, Jones LA, Kahn RS, Kirov G, Landen M, Leboyer M, Lewis CM, Li QS, Lissowska J, Martin NG, Mayoral F, McElroy SL, McIntosh AM, McMahon FJ, Melle I, Metspalu A, Mitchell PB, Morken G, Mors O, Mortensen PB, Muller-Myhsok B, Myers RM, Neale BM, Nimgaonkar V, Nordentoft M, Nothen MM, O'Donovan MC, Oedegaard KJ, Owen MJ, Paciga SA, Pato C, Pato MT, Posthuma D, Ramos-Quiroga JA, Ribases M, Rietschel M, Rouleau GA, Schalling M, Schofield PR, Schulze TG, Serretti A, Smoller JW, Stefansson H, Stefansson K, Stordal E, Sullivan PF, Turecki G, Vaaler AE, Vieta E, Vincent JB, Werge T, Nurnberger JI, Wray NR, Di Florio A, Edenberg HJ, Cichon S, Ophoff RA, Scott LJ, Andreassen OA, Kelsoe J, Sklar P; Bipolar Disorder Working Group of the Psychiatric Genomics Consortium. Genome-wide association study identifies 30 loci associated with bipolar disorder. Nat Genet. 2019 May;51(5):793-803. doi: 10.1038/s41588-019-0397-8. Epub 2019 May 1. PMID 31043756
- See also: Related Info — https://www.neuropsybit.org/data-governance
- See also: Related Info — https://www.neuropsybit.org
- See also: Related Info — https://www.rtsgd.org
- Available data/document: "De-identified clinical, phenotypic, Genotypic Raw, and biospecimen metadata; laboratory quality control metrics; and data dictionaries describing collected variables — https://www.neuropsybit.org/data-governance